CLINICAL TRIAL: NCT02557165
Title: Impact of Chronic Obstructive Pulmonary Disease on Peripheral and Respiratory Muscle Regeneration
Brief Title: Impact of COPD on Muscle Regeneration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: CRT114804
Record Dates: First submitted 2015-09-02; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: COPD
Keywords: Muscle regeneration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscle biopsies from the quadriceps and diaphragm muscles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients: Patients with mild to moderate COPD having a scheduled lung surgery. Vastus lateralis and diaphragm muscle biopsies performed during surgery
  Interventions: Procedure: Muscle biopsies
- Patients with normal lung function: Patients with normal lung function having a scheduled lung surgery. Vastus lateralis and diaphragm muscle biopsies performed during surgery.
  Interventions: Procedure: Muscle biopsies

INTERVENTIONS:
Procedure: Muscle biopsies — Muscle biopsies will allow acces to samples for observational studies. Vastus latetalis: needle biopsy (Bergstrom technique). Diaphragm: open biopsy performed by thoracic surgeon during lung surgery.

SUMMARY:
Muscle weakness and atrophy are important consequences of chronic obstructive pulmonary disease (COPD) and can affect both respiratory and peripheral muscles. Impaired muscle regeneration is thought to be implicated in the process of muscle atrophy. In this study the investigators will evaluate muscle regenerative potential of the Vastus Lateralis (VL) and diaphragm of patients with COPD, compared to patients with normal lung function.

DETAILED DESCRIPTION:
Preliminary results suggest that the activation and differentiation processes of satellite cells isolated from the VL of patients with COPD could be altered. The investigators propose to compare the regenerative potential of the VL and the diaphragm in 15 patients with COPD and 15 individuals with normal lung function undergoing a thoracic surgery. From muscle biopsies, satellite cells will be isolated and cultured to assess their proliferation and differentiation rates, and the expression level of myogenic effectors (MyoD, Myf5, myogenin, and MRF4). Alterations in these measurements will confirm the hypotheses that the regenerative potential is lower in both muscle groups in patients with COPD compared to controls and that in COPD, the regenerative potential is lower in VL compared to the diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a scheduled thoracic surgery
* ≥ 40 years
* Smoking cessation ≥ 1 month
* Smoking history ≥ 10 pack-year

Exclusion Criteria:

* Subjects who received either chemiotherapy or radiotherapy
* Hypoxemia
* Body weight loss ≥ 10%
* Use of systemic corticosteroid in the last month

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a scheduled thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Muscle satellite cell proliferation index | Sequential analyses performed over a period of 2 weeks after tissue collection.
  Isolation from muscle biopsies of satellite cell to evaluate their regeneration capacity by evaluating the proliferation capacity
Muscle satellite cell differentiation index | Sequential analyses performed over a period of 2 months after tissue collection.
  Isolation from muscle biopsies of satellite cell to evaluate their regeneration capacity by evaluating the differentiation capacity

CONTACTS AND LOCATIONS:
Overall Officials: Richard Debigare, PhD, PT, Principal Investigator — Laval University

REFERENCES:
- [Background] Theriault ME, Pare ME, Lemire BB, Maltais F, Debigare R. Regenerative defect in vastus lateralis muscle of patients with chronic obstructive pulmonary disease. Respir Res. 2014 Mar 25;15(1):35. doi: 10.1186/1465-9921-15-35. PMID 24666540
- [Background] Theriault ME, Pare ME, Maltais F, Debigare R. Satellite cells senescence in limb muscle of severe patients with COPD. PLoS One. 2012;7(6):e39124. doi: 10.1371/journal.pone.0039124. Epub 2012 Jun 13. PMID 22720047
- [Background] Caron MA, Debigare R, Dekhuijzen PN, Maltais F. Comparative assessment of the quadriceps and the diaphragm in patients with COPD. J Appl Physiol (1985). 2009 Sep;107(3):952-61. doi: 10.1152/japplphysiol.00194.2009. Epub 2009 Apr 9. PMID 19359618